CLINICAL TRIAL: NCT04551625
Title: Assessment of Colonic Motility in Patients With Diabetes Using High Resolution Colonic Manometry and 3D-Transit.
Brief Title: Colonic Motility in Patients With Diabetes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Aalborg University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HRCM_3DT_DM; EUDRAMED: CIV-20-05-032844 (Other: Danish Medicines Agency)
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Diabetes Mellitus
Keywords: Diabetic enteropathy; Neurogastroenterology; Colonic motility; High Resolution Colonic Manometry; 3D-Transit system
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: High Resolution Colonic Manometry and 3D-Transit system. — Not performed as an intervention, the study is observational.

SUMMARY:
Background:

Gastrointestinal (GI) symptoms are overrepresented in patients with diabetes mellitus (DM) and often have a major impact on quality of life. Typical symptoms of diabetic enteropathy include abdominal pain, nausea, vomiting, diarrhoea, constipation, faecal incontinence, and bloating. Bowel symptoms in DM are usually caused by widespread dysfunction of the GI tract, but the exact pathophysiology remains incompletely understood. Within recent years, new methods for detailed assessment of GI motility have been developed. Hence, the electromagnetic 3D-Transit system is a safe, non-invasive method for detailed description of GI motility. The system tracks the exact position of an ingested electromagnetic capsule through the entire GI tract and provides detailed information on both regional transit- and contraction patterns. High Resolution Colonic Manometry (HRCM) allows extremely detailed description of contraction patterns in the colon. The HRCM is however an invasive method, as the catheter is placed during colonoscopy. HRCM has not previously been performed on diabetic patients and 3D-Transit has only been used sparingly.

Study Objectives:

The purpose of this study is to obtain detailed description of colonic contractions in patients with DM and gastrointestinal symptoms, especially during fast and after meals.

Hypothesis:

1. Patients with DM and GI symptoms have reduced high-amplitude, antegrade contractions in the colon when compared to healthy controls (HRCM).
2. Patients with DM and GI symptoms have reduced long, fast mass-movements when compared to healthy controls (3D-Transit).
3. The contractile response to a meal is reduced in patients with symptoms of diabetic enteropathy when compared to healthy controls.

Materials and methods:

20 patients with DM type 1 or 2 and GI symptoms will be investigated simultaneously HCRM and the 3D-Transit capsule. Data will be compared to the healthy from another study (CIV-19-05-028726). A colonoscopy is performed to install the HRCM catheter and place two 3D-Transit capsules within the colon. For 24 hours, the participants lie in a bed in the research lab while pressure changes from the HRCM catheter are recorded and the 3D-Transit capsules are followed through the gastrointestinal system.

Perspectives:

The study will add to the very limited data available on colonic dysfunction in DM.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or 2 diabetes (at least 3 years since diagnosis)
* Age between 18 and 70
* Gastrointestinal symptoms with a weighted and combined symptomscore >2,3 (assessed with The Gastrointestinal Symptom Rating Scale and The Gastroparesis Cardinal Symptom Score).
* Psychologically able to give an informed content.

Exclusion Criteria:

* Known gastrointestinal disease
* Intake of medication with known effects on the motility patterns in the gastrointestinal system.
* Dysregulated hyperthyroidism or hypothyroidism.
* Any disease known to cause gastroparesis (Parkinson's disease, scleroderma, etc.)
* Pacemaker/ICD
* A scheduled MRI scan within 4 weeks after trial initiation.
* Abdominal circumference >140cm
* Pregnancy and lactation
* Unable to follow the scheduled program in the trial due to mental illness or instability.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All individuals who meet the inclusion- and exclusion criteria can be enrolled in the study. The recruitment process will primarily take place through the outpatient clinics at Aarhus University Hospital.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-10-15 (Estimated); Primary Completion 2022-10-15 (Estimated); Study Completion 2022-10-15 (Estimated)

PRIMARY OUTCOMES:
High amplitude, antegrade contractions assessed with HRCM | All 24 hours of HRCM and 3D-Transit recording
  Quantity, amplitude and duration of the high amplitude, antegrade propagating contractions accessed with HRCM, when compared to healthy controls.

SECONDARY OUTCOMES:
Long, fast mass-movements assessed with 3D-Transit | All 24 hours of HRCM and 3D-Transit recording.
  Quantity and length of the long, fast mass-movements assessed with 3D-Transit, when compared to healthy controls.
Distance of capsule movement. | All 24 hours of HRCM and 3D-Transit recording.
  How do the length of a pressure change measured by HRCM correlate with the distance covered in long fast antegrade movements determined with the 3D-Transit system (cm).

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Krogh, MD, ph.d., Study Chair — Overall scientific leadership of the protocol
Locations (1):
- The Department og Hepatology and gastroenterology, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No